CLINICAL TRIAL: NCT00592761
Title: Treatment of Dysphagia Using the Mendelsohn Maneuver
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R03DC004942 (NIH); R03DC004942 (NIH)
Record Dates: First submitted 2007-12-27; First posted 2008-01-14 (Estimated); Results first posted 2010-07-20 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: Stroke; Dysphagia
Keywords: Deglutition Disorders; Mendelsohn Maneuver; SEMG
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Within subjects treatment, no-treatment (Experimental): Within subject, treatment and no-treatment periods. Each participant served as his/her own control in this AABB/BBAA alternating treatment conditions design. Results were also compared across groups (treatment v. no-treatment).
  Interventions: Behavioral: Mendelsohn Maneuver

INTERVENTIONS:
Behavioral: Mendelsohn Maneuver — Mendelsohn Maneuver with Surface Electromyography

SUMMARY:
The primary goal of the investigation is to determine the effects of the Mendelsohn maneuver on the physiology of the swallow in individuals who have suffered a stroke and exhibit signs of pharyngeal dysphagia.

DETAILED DESCRIPTION:
The primary goal of the investigation is to determine the effects of the Mendelsohn maneuver (voluntary prolongation of laryngeal excursion at the midpoint of the swallow) on the physiology of the swallow in individuals who have suffered a stroke and exhibit signs of pharyngeal dysphagia (specifically, reduced duration of hyoid maximum elevation, reduced extent of hyoid maximum elevation, reduced duration of hyoid maximum anterior excursion, reduced extent of hyoid maximum anterior excursion, and reduced duration of upper esophageal sphincter (UES) opening with subsequent residue in the pyriform sinuses and, potentially, aspiration). Participants are assessed with videofluoroscopy at the initiation of the study and after each week of the study. After the 4 weeks of participation are complete, all participants will be discharged from treatment and will be brought back to the clinic for a final Videofluoroscopic Swallow Study (VFSS) evaluation after 2 weeks. This means that individuals in Group 1 will be re-analyzed after 1 month of additional no-treatment, and Group 2 will be re-analyzed after 2 additional weeks of no-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stroke (1-18 months post)
* Pharyngeal Dysphagia

Exclusion Criteria:

* Other neurologic or structural abnormality to oropharynx
* History of dysphagia prior to latest stroke

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary H McCullough, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- UArkansas/UAMS Medical Center, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of participants occurred through The University of Arkansas for Medical Sciences Medical Center Speech Pathology Clinic and newspaper advertisements between February 2003 and February 2010.
Pre-assignment Details: Participants were only assigned to a group after their initial evaluation and no exclusions were necessary. Participants were each assigned to receive 2 weeks of treatment and two weeks of no treatment. Assignments were randomized so half began with treatment and half began with no treatment.
Groups:
- No Treatment Then Treatment: Participants received 2 weeks of no-treatment and then 2 weeks of treatment with the Mendelsohn manuever.
- Treatment Then No Treatment: Participants received 2 weeks of treatment with the Mendelsohn manuever and then 2 weeks of no treatment.
Period: First Intervention (2 Weeks)
Arm/Group | No Treatment Then Treatment | Treatment Then No Treatment
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | No Treatment Then Treatment | Treatment Then No Treatment
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: This includes all participants. Half received treatment then no treatment and have received no treatment then treatment.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants] — Participants were analyzed for age effects within analysis of variance.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 7
    >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants] — Gender effects were analyzed within the analysis of variance.
  Participants
    Female | 7
    Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Duration of Superior Hyolaryngeal Movement
Description: Change in duration of superior elevation of hyoid bone.
Time Frame: baseline and six weeks
Population: per protocol
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment Then Treatment | Treatment Then No Treatment
Number analyzed (Participants) | 18 | 18
seconds | .213 (.154) | .233 (.184)

2. Secondary Outcome: Change in Oral Intake Ability
Description: Oral Intake Ability was measure with the Dysphagia Outcome and Severity Scale. A 7 is normal and a 1 is complete inability to consume any food safely. The means reported for treatment and no treatment periods are mean changes in scores throughout the period.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Treatment Then Treatment | Treatment Then No Treatment
Number analyzed (Participants) | 18 | 18
units on a scale | 1.8 (.15) | 2.3 (.11)

3. Secondary Outcome: Change in Duration of Opening of Upper Esophageal Sphincter
Description: Change in duration of pre- and post-treatment duration of UES opening.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment Then Treatment | Treatment Then No Treatment
Number analyzed (Participants) | 18 | 18
seconds | .584 (.159) | .610 (.183)

4. Primary Outcome: Change in Duration of Hyoid Maximum Anterior Excursion
Description: Change in the duration of maximum anterior movement of the hyoid bone during swallowing.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment Then Treatment | Treatment Then No Treatment
Number analyzed (Participants) | 18 | 18
seconds | .233 (.157) | .247 (.161)

ADVERSE EVENTS:
Time Frame: Subjects were followed for up to one year after study completion.
Arm/Group | No Treatment Then Treatment | Treatment Then No Treatment
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes